CLINICAL TRIAL: NCT05150093
Title: Deep Brain Stimulation in Laryngeal Dystonia and Voice Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Massachusetts General Hospital (Other); University of Utah (Other); University of California, San Francisco (Other); UMass Memorial Health (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Kristina Simonyan, Professor of Otolaryngology - Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P003236
Record Dates: First submitted 2021-11-27; First posted 2021-12-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Laryngeal Dystonia; Spasmodic Dysphonia; Tremor; Dystonia
MeSH Terms: conditions — Dysphonia; Tremor; Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrophysiological signal data collection (Experimental): Patients diagnosed with dystonia or tremor who are recommended for DBS surgery. Electrophysiological data will be collected at the time of DBS surgery.
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Clinically indicated DBS treatment for dystonia or tremor with simultaneous research electrocorticography (ECoG).

SUMMARY:
The goals of this project are 1) to determine the incidence of neurological voice disorders in patients with dystonia and essential tremor undergoing deep brain stimulation (DBS), 2) investigate the neuroimaging and intracranial neurophysiology correlates of voice dysfunction in these subjects, and subsequently 3) determine the effects of DBS on voice function.

DETAILED DESCRIPTION:
Loss of voice control, which is critical for conveying effective spoken communication, is often a significant feature in patients with movement disorders, such as dystonia and essential tremor. Voice dysfunction, however, has been overshadowed clinically by a focus on limb motor symptoms. For example, deep brain stimulation (DBS) effectively reduces limb dystonia and tremor in these patients, but the modulation of voice symptoms by DBS has been vastly understudied. It is assumed that the production and modulation of voice are regulated by the basal ganglia-thalamo-cortical network in a loop architecture that is common to all motor behaviors. There is, however, little empirical data to inform our specific understanding of how voice function is encoded in basal ganglia-thalamo-cortical interactions. The overall goal of this research is to use a combination of invasive and non-invasive human neuroscience to improve our understanding of the incidence and neural correlates of neurological voice disorders (laryngeal dystonia and voice tremor) in patients with isolated dystonia and essential tremor undergoing DBS surgery. The investigators will use simultaneous electrocorticography (ECoG) and subcortical activity recording in dystonia and tremor patients who are awake and speaking during DBS implantation surgery. The results of this research will inform the development of strategies for closed-loop brain stimulation specifically to treat neurological voice dysfunction that can be tested in a subsequent clinical trial.

ELIGIBILITY:
Inclusion

1. Clinical indications to proceed with DBS implantation, as determined by the clinical multidisciplinary movement disorders board, including: a) definitive diagnosis of essential tremor or dystonia, b) medically refractory disease, c) adequate performance on neuropsychological evaluation as determined by a licensed clinical neuropsychologist.
2. The ability to comply with test directions, complete pre-operative task training, and provide informed consent.
3. Age 18-80 years.

Exclusion

1. Inability to understand or perform the task outlined in the protocol during a pre-surgery training session. 2. Significant hearing loss.

3. Cortical venous anatomy that could potentially obstruct ECoG electrode placement, as determined by the surgeon, visualized on pre-op MRI or during surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Correlations between brain signals and intraoperative voice and speech production performance. | 5 years
  Analysis of intraoperative recordings from deep basal ganglia structures and cortical regions relevant to voice and speech control.
Changes in standard clinical outcome for dystonia patients | 5 years
  Quantitative measures of voice and motor changes following deep brain stimulation surgery using standard clinical criterion of Burk-Fahn-Marsden Dystonia Rating Scale where higher score means a worse outcome.
Changes in standard clinical outcome for tremor patients | 5 years
  Quantitative measures of voice and motor changes following deep brain stimulation surgery using standard clinical criterion of Fahn-Tolosa-Marin Tremor Rating Scale where higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Study Director — Massachusetts Eye and Ear
Locations (1):
- Massachusetts General Hospital, University of California San Francisco, University of Utah, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No